CLINICAL TRIAL: NCT00383045
Title: HIV Risk Reduction and Drug Abuse Treatment in Malaysia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0103012336; R01DA014718-04 (NIH)
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2009-02

CONDITIONS: Opiate Dependence
Keywords: Buprenorphine; Naltrexone; HIV risk reduction behavior; Counseling
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Naltrexone

INTERVENTIONS:
Drug: Buprenorphine/Subutex
Drug: Naltrexone
Procedure: Drug counseling

SUMMARY:
A randomized clinical trial comparing drug abuse and HIV risk reduction counseling (DC-HIV) alone, DC-HIV combined with naltrexone maintenance, and DC-HIV combined with buprenorphine maintenance for the treatment of heroin addicts in Malaysia.

DETAILED DESCRIPTION:
Combining drug abuse and HIV risk reduction counseling with opioid agonist maintenance treatment (OMT) or antagonist maintenance treatment with naltrexone (NMT) is effective for reducing illicit drug use and preventing HIV transmission associated with heroin dependence, but support for NMT and OMT remains tenuous in many Western Pacific countries (e.g., Malaysia, Indonesia and Singapore) where heroin addiction and HIV infection are epidemic and closely linked due to injection drug use (IDU) and high-risk sexual behaviors among addicts. Promising results of NMT in Malaysia have created interest in evaluating OMT using buprenorphine (BMT) and comparing the efficacy of counseling alone and counseling combined with BMT or NMT. This 24-week, randomized double blind clinical trial compares the efficacy for preventing heroin use and relapse and reducing HIV risk behaviors of manual-guided, HIV risk reduction and drug counseling (DC-HIV) alone or when combined with buprenorphine maintenance treatment (BMT) or naltrexone maintenance treatment (NMT) for recently detoxified and currently abstinent heroin dependent patients (N=180) in Malaysia (Specific Aim 1). The study will allow evaluation of 3 hypotheses: DC-HIV plus naltrexone is superior to DC-HIV alone; DC-HIV plus buprenorphine is superior to DC-HIV alone; and DC-HIV plus naltrexone is superior to DC-HIV plus buprenorphine. Primary outcome measures, assessed by 3x/wk urine toxicology testing and self-report, include resumption of heroin use, 1 or 3 weeks continuous relapse and reductions in HIV risk behaviors. The project will also evaluate the characteristics of treatment-seeking heroin addicts in Malaysia (including specific risk behaviors and patterns of HIV risk behaviors; prevalence of psychiatric and other medical comorbidity; and patterns of social, family, vocational, and criminal activity and service needs-Specific Aim 2). This data will be used to revise the DC-HIV manual to address the specific circumstances and risk behaviors of Malaysian heroin addicts. Finally, the project provides clinical training for health professionals and training and mentoring in drug abuse treatment and HIV prevention research to clinical researchers who will continue development, implementation, evaluation and dissemination of HIV prevention and drug abuse treatment approaches in Malaysia after the project ends (Specific Aim 3). The results of the study will inform government policy and support for HIV prevention and drug abuse treatment efforts in Malaysia and possibly also in other Western Pacific countries.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependence

Exclusion Criteria:

* Dependence on alcohol, benzodiazepines or sedatives
* Suicide or homicide risk
* Psychotic disorder or major depression
* Inability to read or understand the protocol or assessment questions
* Life-threatening or unstable medical problems
* Greater than 3 times normal liver enzymes (AST, GGT)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to resumption of heroin use
Time to relapse
Maximum consecutive weeks of opiate abstinence
Reduction of HIV risks

SECONDARY OUTCOMES:
Addiction-related functional status
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Schottenfeld, M.D., Principal Investigator — Yale University; Mahmud Mazlan, M.D., Study Director — Hospital Muar, Malaysia
Locations (2):
- Yale University School of Medicine, New Haven, Connecticut, United States
- Substance Abuse Research Center, Muar town, Johor, Malaysia

REFERENCES:
- [Background] Mazlan M, Schottenfeld RS, Chawarski MC. New challenges and opportunities in managing substance abuse in Malaysia. Drug Alcohol Rev. 2006 Sep;25(5):473-8. doi: 10.1080/09595230600883354. PMID 16939945
- [Background] Chawarski MC, Mazlan M, Schottenfeld RS. Heroin dependence and HIV infection in Malaysia. Drug Alcohol Depend. 2006 Apr;82 Suppl 1:S39-42. doi: 10.1016/s0376-8716(06)80007-4. PMID 16769444
- [Derived] Schottenfeld RS, Chawarski MC, Mazlan M. Maintenance treatment with buprenorphine and naltrexone for heroin dependence in Malaysia: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Jun 28;371(9631):2192-200. doi: 10.1016/S0140-6736(08)60954-X. PMID 18586174